CLINICAL TRIAL: NCT04554706
Title: Using Mobile Phones to Reduce Negative Rumination
Brief Title: Evaluating a Mobile Phone Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Lynn Miller, Professor of Communication, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: UscCalifornia
Record Dates: First submitted 2020-06-26; First posted 2020-09-18 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Depression; Rumination - Thoughts
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: There are three conditions: a JITAI interactive narrative condition, a JITAI non-narrative condition, and a wait-list control condition.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant blind to condition assigned to (compared to alternatives), assignment is automatic/random via computer so investigator blind to participant assignment; analyst is blind to meaning of condition codes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- a JITAI interactive narrative condition (Narrative JITAI) (Experimental): This arm is an exploratory condition, which tested whether story-based JITAI would be an effective way to deal with rumination.
  Interventions: Behavioral: Mobile-phone delivered Treatment for Excessive Rumination
- a JITIAI non-interactive condition (Experimental): This arm uses the regular JITAI ( mobile phone delivered) intervention to provide treatment for ruminative thoughts.
  Interventions: Behavioral: Mobile-phone delivered Treatment for Excessive Rumination
- a wait-list control condition (No Intervention): Participants in this arm will be put on a waitlist without receiving active treatment upon the end of the study.

INTERVENTIONS:
Behavioral: Mobile-phone delivered Treatment for Excessive Rumination — This is a one-month three-arm clinical control trial to reduce the rumination and interpersonal impairment link.
  Arms: a JITAI interactive narrative condition (Narrative JITAI); a JITIAI non-interactive condition

SUMMARY:
This clinical trial intends to study the efficacy of a mobile phone delivered intervention in reducing depression-related rumination.

DETAILED DESCRIPTION:
Here we propose to test a novel intervention to help individuals manage their depressive rumination. The intervention is based on a just-in-time, adaptive-intervention (JITAI) design. A JITAI is "an intervention designed to address the dynamically changing needs of individuals via the provision of the type/amount of support needed, at the right time, and only when needed ." This study is also to address one major concern regarding designing JITAI interventions: the burden on participants in having to be engaged with the intervention through diaries, self-reports, and other forms of assessment procedures daily. To reduce this burden, we first pilot test an interactive narrative form. An interactive narrative is an essential form of storytelling that involves certain interactive features such that audiences or readers of the story can have the feeling that they are actively engaging in certain forms of interactions with the story characters.

To test the efficacy of such an intervention, there will be a one-month three-arm clinical control trial to reduce depressive rumination. There are three conditions: a JITAI interactive narrative condition, a non-narrative JTIAI condition, and a wait-list control condition. This study could contribute to our knowledge in designing more effective interventions in curbing depression using mobile technology. It can also advance our theoretical knowledge of the role of interactive narratives in reducing user burden in mobile health.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a current self-reported clinical diagnosis of being depressed ( mild to moderate depression and major depressive disorder)
* Participants should be 18 or older.
* Participants should have a working smartphone and daily access to the internet.

Exclusion Criteria:

-Participants who do not have regular access to the internet and a smart phones will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-11-06 (Actual); Study Completion 2021-11-06 (Actual)

PRIMARY OUTCOMES:
Change in Rumination focus ( immediately after intervention) | Change in Rumination focus at the baseline and immediate-post intervention (measured baseline, immediate-post intervention, and two-week follow-up).
  Momentary Ruminative Self-Focus Inventory-Abbreviated (MRSI-A). The MRSI is a 6-item questionnaire measuring state-level fluctuations in ruminative self-focus. Each item ranges from 1 (Strongly disagree) to 7 (Strongly agree).
Change in Rumination focus ( two weeks after intervention) | Change in Rumination focus at the baseline and two weeks after the intervention (measured baseline, immediate-post intervention, and two-week follow-up).
  Momentary Ruminative Self-Focus Inventory-Abbreviated (MRSI-A). The MRSI is a 6-item questionnaire measuring state-level fluctuations in ruminative self-focus. Each item ranges from 1 (Strongly disagree) to 7 (Strongly agree).
Change in Heart-rate( baseline and immediately after intervention) | Change in heart rates at the baseline and immediate-post intervention .(measured baseline, immediate-post intervention, and two-week follow-up)
  Participants self-report their heart-rate by using a moblie phone app by the name of Instant Heart rate (see example outcome report: https://www.azumio.com/heartrate/report.jsp?token=28928192047-28935807244-3eb659-334dc9f600fc7084f8cda95b135396673b2bd118-1588095873083#)
Change in Heart-rate (baseline and two weeks after intervention.) | Change in heart rates at the baseline and two weeks after the intervention (measured baseline, immediate-post intervention, and two-week follow-up).
  Participants self-report their heart-rate by using a moblie phone app by the name of Instant Heart rate (see example outcome report: https://www.azumio.com/heartrate/report.jsp?token=28928192047-28935807244-3eb659-334dc9f600fc7084f8cda95b135396673b2bd118-1588095873083#)
Change in Depressive Symptoms ( baseline and immediately after intervention) | Change in depressive symptoms at the baseline and immediate-post intervention .(measured baseline, immediate-post intervention, and two-week follow-up)
  a 3-item scale in which participants rated their level of depressed mood, anhedonia, and irritability on 7-point Likert scales ranging from 1 (Not at all) to 7 (Very much) at the time of the alert. The SDS is in part modeled after a scale used in a previous EMA study of rumination and depression (Moberly & Watkins, 2008a). The scale was presented as a slider bar on participants' smartphones."
Change in Depressive Symptoms (baseline and two weeks after intervention.) | Change in depressive symptoms at the baseline and two weeks after the intervention (measured baseline, immediate-post intervention, and two-week follow-up).
  a 3-item scale in which participants rated their level of depressed mood, anhedonia, and irritability on 7-point Likert scales ranging from 1 (Not at all) to 7 (Very much) at the time of the alert. The SDS is in part modeled after a scale used in a previous EMA study of rumination and depression (Moberly & Watkins, 2008a). The scale was presented as a slider bar on participants' smartphones."

OTHER OUTCOMES:
Change in Ruminative symptom ( baseline and immediately after intervention) | Change in ruminative symptoms at the baseline and two weeks after the intervention (measured baseline, immediate-post intervention, and two-week follow-up).
  To measure this, we will use the ruminative response scale (RRS), a self-report measure of describing one's responses to depressed mood. It has 22 items, ranging from 1 (not like me at all) to 7 (A lot like me).
Change in Ruminative symptom (baseline and two weeks after intervention.) | Change in ruminative symptoms at the baseline and two weeks after the intervention (measured baseline, immediate-post intervention, and two-week follow-up).
  To measure this, we will use the ruminative response scale (RRS), a self-report measure of describing one's responses to depressed mood. It has 22 items, ranging from 1 (not like me at all) to 7 (A lot like me).

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Miller, Ph.D, Principal Investigator — UscCalifornia
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Because this study is a pilot study, we decided not to share the data.

REFERENCES:
- [Background] Nahum-Shani I, Hekler EB, Spruijt-Metz D. Building health behavior models to guide the development of just-in-time adaptive interventions: A pragmatic framework. Health Psychol. 2015 Dec;34S(0):1209-19. doi: 10.1037/hea0000306. PMID 26651462
- [Background] Sharmin M, Raij A, Epstien D, Nahum-Shani I, Beck JG, Vhaduri S, Preston K, Kumar S. Visualization of Time-Series Sensor Data to Inform the Design of Just-In-Time Adaptive Stress Interventions. Proc ACM Int Conf Ubiquitous Comput. 2015 Sep;2015:505-516. doi: 10.1145/2750858.2807537. PMID 26539566
- [Background] Walter N, Murphy ST, Frank LB, Baezconde-Garbanati L. Each Medium Tells a Different Story: The Effect of Message Channel on Narrative Persuasion. Commun Res Rep. 2017;34(2):161-170. doi: 10.1080/08824096.2017.1286471. Epub 2017 Mar 2. PMID 30739986
- [Derived] Wang L, Miller L. Assessment and Disruption of Ruminative Episodes to Enhance Mobile Cognitive Behavioral Therapy Just-in-Time Adaptive Interventions in Clinical Depression: Pilot Randomized Controlled Trial. JMIR Form Res. 2023 Jan 5;7:e37270. doi: 10.2196/37270. PMID 36602841